CLINICAL TRIAL: NCT03603652
Title: A Multicenter Study of the NEUWAVE Flex Microwave Ablation System in the Ablation of Medically Inoperable Primary Soft Tissue Lesions of the Lung: An Initial Experience
Brief Title: NEUWAVE Flex Microwave Ablation System in the Ablation of Primary Soft Tissue Lesions of the Lung
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study originally suspended pending a protocol amendment but study now terminated.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2017_06
Record Dates: First submitted 2018-05-16; First posted 2018-07-27 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma
Keywords: Lung Lesions; Soft Tissue- Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microwave Ablation (Experimental): Ablations will be performed under general anesthesia via transbronchial approach by an interventional pulmonologist or thoracic surgeon.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — Ablations will be performed under general anesthesia via transbronchial approach by an interventional pulmonologist or thoracic surgeon. Prior to the ablation, the treating physician will perform an endobronchial ultrasound to confirm disease staging.

SUMMARY:
Patients with medically inoperable primary soft tissue lesion of the lung will have transbronchial microwave ablation performed via transbronchial approach by an interventional pulmonologist or thoracic surgeon using CT imaging. Prior to the ablation procedure, the treating physician will use endobronchial ultrasound to confirm staging. Patients will be followed for one year following the ablation procedure for efficacy and safety.

DETAILED DESCRIPTION:
Patients with medically inoperable primary soft tissue lesion of the lung (lesions less than or equal to 2cm and located in the outer two-thirds of the lung and not closer than 1cm to the pleura) will have transbronchial microwave ablation performed using CT imaging. All ablations will be performed under general anesthesia via transbronchial approach by an interventional pulmonologist or thoracic surgeon.

Prior to the ablation procedure, the treating physician will use endobronchial ultrasound to confirm staging.

Patients will be followed for one year following the ablation procedure for efficacy and safety with specific follow-up visits at 30 days, 6 months, and 12 months post-ablation. A user experience questionnaire is completed by the treating physician to better understand the ease of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Patients ≥ 18 years old.
3. Performance status 0-2 via ECOG (Eastern Cooperative Oncology Group) classification.
4. Willing to fulfill all follow-up visit requirements.
5. Medically inoperable primary soft tissue lesion of the lung or patient election not to have surgery. (Medically inoperable is defined per the following indicators: post op predictive FEV1 (forced expiratory volume in 1 second) < 40%; DLCO (diffusing capacity of the lung for carbon monoxide) < 40%; hypoxemia or hypercapnia diabetes with end-organ damage; or severe cerebral, cardiovascular, peripheral vascular disease, or chronic heart disease)
6. One soft tissue lesion ≤ 2 cm in the outer two thirds of the lung and not closer than 1 cm to the pleura.

   (Outer two thirds of the lung is defined as peripheral beyond the segmental airway, past the segmental bronchi, such that proximal endobronchial soft tissue lesions are avoided; soft tissue lesions should not be contiguous with the pleura)
7. Radiographic resolution of pneumonia

Exclusion Criteria:

1. Scheduled concurrent procedure for the target soft tissue lesion other than those that are lung related.
2. Pregnant or breastfeeding.
3. Physical or psychological condition that would impair study participation.
4. Patients with uncorrectable coagulography at time of screening.
5. Patient with implantable devices, including pacemakers or other electronic implants.
6. Prior pneumonectomy or bronchiectasis.
7. Severe neuromuscular disease.
8. Platelet count ≤ 50,000/mm3.
9. ASA (American Society of Anesthesiologists) score of ≥ 4.
10. Inability to tolerate anesthesia.
11. Expected survival less than 6 months.
12. Clinically significant hypertension.
13. Chronic ventilator support, which uses bi-level positive airway pressure (PAP).
14. Endobronchial soft tissue lesions proximal to the segmental airways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gildea, MD, Principal Investigator — The Cleveland Clinic; Michael Pritchett, MD, Principal Investigator — FirstHealth Moore Regional Hospital; Janani Reisenauer, MD, Principal Investigator — Mayo Clinic; Bradley Pua, MD, Principal Investigator — Cornell; Jae Kim, MD, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian-Weill Cornell Medicine, New York, New York
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Microwave Ablation: Each participant underwent microwave ablation to the original soft tissue lesion in the lung at single visit. The treating physician determined the ablation time and power used on a case-by-case basis.
Period: Overall Study
Arm/Group | Microwave Ablation
Started | 10
Completed | 8
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: 10 patients were enrolled and treated
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of patient at the time they signed the Informed Consent Form.
  Years | 69.3 (7.689)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI)
  kg/m^2 | 26.8 (4.469)
Smoking Status [Count of Participants; unit: Participants] — Patients who were current smokers, former smokers, or non-smokers.
  Participants
    Current Smoker | 3
    Former Smoker | 6
    Non-Smoker | 1
Radiation History [Count of Participants; unit: Participants]
  Yes, radiation history | 1
  No, radiation history | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Ablation Resulted in Technical Success
Description: Ablation of the target lesion according to the protocol and covered completely, with an adequate margin, as defined by the performing physician (that is, the ablation zone completely overlaps or encompasses the target lesion plus an ablative margin), as assessed by CBCT imaging, immediately following the procedure.
Time Frame: Immediately post-ablation (day 0)
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Participants
  10 | 10

2. Primary Outcome: Number of Patients Whose Ablation Resulted in Technique Efficacy
Description: Ablation of the target lesion according to the protocol and covered completely, with an adequate margin, as defined by the performing physician (that is, the ablation zone completely overlaps or encompasses the target lesion plus an ablative margin), as assessed by CT imaging, 30 days (+/- 7 days) after the first ablation procedure.
Time Frame: 30 days post-ablation
Population: Patients analyzed at 30 days post-ablation.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Number of Patients Who Experienced Target Lesion Recurrence
Description: Analyzed at 6 months and 1 year post-ablation via CT imaging
Time Frame: measured at 6 months and 1 year post-ablation
Population: Only 9 patients were analyzed at 6 months post-ablation as 1 patient passed away before the 6 month study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Number of Patients Who Were Readmitted to the Hospital
Description: Any readmission to the hospital within 30 days of the ablation procedure.
Time Frame: Within 30 days post-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Participants | 1

5. Primary Outcome: User Experience Survey (Part I)
Description: A Sponsor-created survey completed by the treating physician immediately post-ablation. Questions were all YES/NO.
Time Frame: Immediately post-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Participants
  Probe through channel as expected: YES | 10
  Probe repositioned after first ablation: YES | 6
  Ablation with NeuWave is predictable: YES | 10
  Ablation with FLEX is simple to use: YES | 10
  Success achieved similar to perc.: YES | 10
  Locate probe/lesion with imaging: YES | 10
  Locate ablation zone created: YES | 7

6. Primary Outcome: User Experience Survey (Part II)
Description: A Sponsor-created survey completed by the treating physician immediately post-ablation. This question asked the time it took to place the probe in a position that was ready for ablation.
Time Frame: Immediately post-ablation
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Minutes | 18.2 (11.25)

7. Primary Outcome: User Experience Survey (Part III)
Description: A Sponsor-created survey completed by the treating physician immediately post-ablation. This question asked how many cone-beam CT (CBCT) scans were taken to place the probe such that it was ready for ablation.
Time Frame: Immediately post-ablation
Measure: Mean (Standard Deviation); unit: Count of Scans
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Count of Scans | 4.4 (3.44)

8. Primary Outcome: User Experience Survey (Part IV)
Description: A Sponsor-created survey completed by the treating physician immediately post-ablation. This question asked the distance of the tip of the probe to the center of the soft-tissue lesion (in mm) just before the ablation procedure was initiated.
Time Frame: Immediately post-ablation
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Millimeters | 4.1 (2.23)

9. Primary Outcome: User Experience Survey (Part V)
Description: A Sponsor-created survey completed by the treating physician immediately post-ablation. This question asked how many times the probe had to be repositioned to complete the ablation procedure.
Time Frame: Immediately post-ablation
Measure: Mean (Standard Deviation); unit: Count of Probe Repositions
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 10
Count of Probe Repositions | 0.9 (0.93)

ADVERSE EVENTS:
Time Frame: 1 year following the initial ablation procedure.
Description: Participants were evaluated for AEs and SAEs at every study visit starting with the ablation procedure through the end-of-study (1 year following the initial ablation procedure).
Arm/Group | Microwave Ablation
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation (N=10)
Ataxia (Nervous system disorders) | 1 (1) — worsening ataxia symptoms
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (5) — worsening or flare-up of pre-existing condition.
Infected Bite (Infections and infestations) | 1 (1) — cellulitis of the right hand from infected cat bite.
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation (N=10)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03603652/SAP_000.pdf
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03603652/Prot_001.pdf